CLINICAL TRIAL: NCT07045662
Title: Effectiveness of Health Literacy in Patients With Type 2 Diabetes Mellitus on a Primary Health Care Protocol: a Randomized Pragmatic Trial
Brief Title: Health Literacy in Patients With Type 2 Diabetes Mellitus.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ernanda Mezaroba (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Sponsor-Investigator, Ernanda Mezaroba, PhD student, Federal University of Rio Grande do Sul
Organization: Federal University of Rio Grande do Sul (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE 79433824.3.0000.5347
Record Dates: First submitted 2025-04-24; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Health literacy.; Type 2 Diabetes Mellitus.; Health education.; Primary health care.; Pragmatic clinical trial.
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Assessment (No Intervention): The participants in the usual assessment were provided regular care, including at least one medical appointment every six months with prescription review.
- Multidisciplinary Assessment (Active Comparator): The participants in the multidisciplinary assessment were followed by teams from the study target-units, by individual and collective interviews, which mirror the care protocol. The frequency of individual visits was at least every six months by a nurse, a physician, and a nutritionist. Regarding the collective activities, the educational groups met for approximately 1 hour and 30 minutes on monthly basis over a period of six months. Considering that there were two FHU in the IG, each team held one activity per month. For the development of the collective activities, methods recognized for intensifying integration and participation, such as using simple language and confirming the participants' understanding of the information covered in the group were recommended.
  Interventions: Behavioral: Multidisciplinary Assessment

INTERVENTIONS:
Behavioral: Multidisciplinary Assessment — The participants in the multidisciplinary assessment were followed by multidisciplinary teams from the study target-units, by individual and collective interviews, which mirror the care protocol. The frequency of individual visits was at least every six months by a nurse, a physician, and a nutritionist.
  Regarding the collective activities, the educational groups met for approximately 1 hour and 30 minutes on monthly basis over a period of six months. Considering that there were two FHU in the IG, each team held one activity per month.
  For the development of the collective activities, methods recognized for intensifying integration and participation, such as using simple language and confirming the participants' understanding of the information covered in the group were recommended.
  Arms: Multidisciplinary Assessment

SUMMARY:
The primary objective of this pragmatic trial was to analyze the effectiveness of health literacy in patients with type 2 Diabetes mellitus (DM2) on a protocol of care in Primary Health Care (PHC) units. The secondary objective was to analyze the effectiveness of knowledge about diabetes, self-efficacy, and glycated hemoglobin (HbA1c) in DM2 patients on a PHC protocol, as compared to the regular care provided by the municipality. Patients from four Family Health Units (FHU) were part of the study, two units as control group (CG) - Usual Assessment, two as intervention group (IG) - Multidisciplinary Assessment, with 44 subjects in each group. The IG mirrors the care protocol, which includes individual visits with physician, nurse, and nutritionist, in addition to systematized collective activities. The CG received the usual care. The research raises the hypothesis that subjects in the IG had a better understanding of aspects related to the disease and were more active in their own health care, as compared to patients who did not receive the intervention.

DETAILED DESCRIPTION:
This research was structured together with professionals who work in the management of the Municipal Health Department of the municipality under study due to the intention of implementing multidisciplinary care for people with Diabetes Mellitus, considering health literacy (HL) and national guidelines as the basis for structuring the assessment protocol. The research is also part of the Municipal Government Program, enhancing the knowledge translation and social impact. Therefore, it was decided to carry out a pragmatic trial, characterized by evaluating the effectiveness of interventions in a real scenario (Zuidgeest et al., 2017). The development of pragmatic trials contribute to the identification of scientific evidence that reduces gaps in primary health care, improving the Brazilian public health system.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Type 2 Diabetes mellitus Disease
* Must be able to read and speak Portuguese
* Being followed exclusively at the primary health care unit for the disease at the beginning of the study
* Not participating in other studies involving diabetes mellitus

Exclusion Criteria:

* Pregnancy
* Physical health problems that prevent the patient from coming to the unit
* Hearing impairment that compromises communication
* Cognitive problems according to the MMSE cutoff points
* History of serious psychiatric disorder recorded in the medical record
* Patients not located after three attempts of home visits on different days and times

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2024-07-12 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Health literacy through the use of Health Literacy Questionnaire - HLQ. | From enrollment to the end of treatment at 6 months.
  The HLQ (Osborne et al.,2013) consists of 9 scales representing 9 dimensions of health literacy: Feeling understood and supported by healthcare providers; Having sufficient information to manage my health;Actively managing my health;Social support for health;Appraisal of health information;Ability to actively engage with healthcare providers;Navigating the healthcare system;Ability to find good health information;Understand health information well enough to know what to do.
  Each HLQ scale has 4-6 items. The HLQ does not provide one overall summative score. The scoring of the HLQ is 9 scale scores, calculated by averaging the item scores within each scale with equal weighting. The 9 scale scores will reflect a person's strengths and needs in the different dimensions of health literacy, with higher scores meaning greater health literacy.
  For Scales 1 to 5, the score range is between 1 and 4 (4 response options). For Scales 6 to 9, the score range is between 1 and 5 (5 response options).

SECONDARY OUTCOMES:
Knowledge about diabetes. | From enrollment to the end of treatment at 6 months.
  Knowledge about DM will be measured by the Diabetes Knowledge Scale (DKN-A). The DKN-A, with 15 multiple-choice questions, addresses several aspects related to general knowledge of diabetes, through 5 categories: a) basic physiology, including the action of insulin; b) hypoglycemia; c) food groups and their replacements; d) management of diabetes in the presence of another disease; e) general principles for disease care. The measurement scale is 0-15 and each item has the following score: one (1) for a correct answer and zero (0) for an incorrect answer. Items 1 to 12 require a single correct answer. For questions 13 to 15, two answers are correct and both must be correct to obtain a score of one. A score of 0 to 8 points indicates little knowledge and greater than 8 points indicates good knowledge about diabetes (Dunn et al., 1984).
Diabetes Management Self-efficacy Scale for Patients with Type 2 Diabetes Mellitus | From enrollment to the end of treatment at 6 months.
  Self-efficacy will be assessed using the Diabetes Management Self-efficacy Scale for Patients with Type 2 Diabetes Mellitus (DMSES). The DMSES has 20 items, distributed across four factors (specific nutrition and weight; general nutrition and drug treatment; physical exercise; blood glucose). The scale items describe the behaviors that people with DM should perform for each of the aforementioned care practices and ask whether they feel able to perform these practices (Bijl; Poelgeest-Eeltink; Shortridge-Baggett, 1999). A Likert-type scale is used to respond to each item, with the following response and scoring pattern: definitely yes (5 points); probably yes (4 points); don't know (3 points); probably no (2 points); definitely no (1 point). SE is determined by the overall mean of the instrument: the scores for each item are added together and divided by the number of items. Higher means indicate greater self-efficacy.
Glycosylated Hemoglobin | From enrollment to the end of treatment at 6 months.
  Glycosylated hemoglobin (HbA1c) is a blood test that measures the average blood glucose levels over the last 3 to 4 months and is routinely used to assess glycemic control in people with diabetes. The target HbA1c result for people with diabetes is around 7.0%, however it varies according to age and presence of comorbidities. Higher values indicate that blood glucose levels are not adequate.
Health conditions | From enrollment to the end of treatment at 6 months.
  The health conditions questionnaire includes the following items:
  - Presence of diseases associated with DM: Eye problems Kidney problems Blood circulation problems Foot problems Other
  - Presence of other morbidities: High blood pressure Obesity Chronic kidney disease Heart disease Depression Anxiety disorder Hypothyroidism Hyperthyroidism Fibromyalgia Cancer Asthma Hypercholesterolemia Cartilage/bone inflammation/degeneration Other
  - Smoking: Yes No
  - Use of alcoholic beverages: Yes No
  - Practice of physical activity: Yes No
  - Body mass index: Underweight: BMI less than 18.5 kg/m² Normal weight: BMI between 18.5 and 24.9 kg/m² Overweight: BMI between 25 and 29.9 kg/m² Obesity: defined as a BMI ≥ 30 kg/m²
  - Abdominal circumference (reference values): Women: ≤ 80 cm Men: ≤ 94 cm
  - Number of consultations with nurses, physicians, and nutritionists over the past six months (assessed only in the second data collection phase)

CONTACTS AND LOCATIONS:
Overall Officials: Idiane Rosset, PhD, Study Director — Federal University of Rio Grande do Sul
Locations (1):
- Federal University of Rio Grande do Sul, Porto Alegre, Brazil

IPD SHARING:
Plan to Share IPD: No
At this stage, I do not intend to share the data collected in this study, as it is part of my doctoral thesis and we intend to analyze it for future publication in peer-reviewed scientific journals at first. Moreover, the decision to withhold the data corroborates with the guidelines established by the Research Ethics Committee, which emphasize that such information must remain under the sole responsibility of the researcher.

REFERENCES:
- [Background] Osborne RH, Batterham RW, Elsworth GR, Hawkins M, Buchbinder R. The grounded psychometric development and initial validation of the Health Literacy Questionnaire (HLQ). BMC Public Health. 2013 Jul 16;13:658. doi: 10.1186/1471-2458-13-658. PMID 23855504
- [Background] Dunn SM, Bryson JM, Hoskins PL, Alford JB, Handelsman DJ, Turtle JR. Development of the diabetes knowledge (DKN) scales: forms DKNA, DKNB, and DKNC. Diabetes Care. 1984 Jan-Feb;7(1):36-41. doi: 10.2337/diacare.7.1.36. PMID 6705664
- [Background] Bijl JV, Poelgeest-Eeltink AV, Shortridge-Baggett L. The psychometric properties of the diabetes management self-efficacy scale for patients with type 2 diabetes mellitus. J Adv Nurs. 1999 Aug;30(2):352-9. doi: 10.1046/j.1365-2648.1999.01077.x. PMID 10457237